CLINICAL TRIAL: NCT00903474
Title: Mindful Movement Program for Breast Cancer Survivors
Brief Title: Mindful Movement Program in Improving Quality of Life in Older Female Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 08061; CHNMC-08061
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Anxiety Disorder; Breast Cancer; Cancer Survivor; Cognitive/Functional Effects; Depression; Psychosocial Effects of Cancer and Its Treatment
Keywords: anxiety disorder; depression; cognitive/functional effects; psychosocial effects of cancer and its treatment; cancer survivor; breast cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Depression | interventions — Exercise Therapy; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: CAM exercise therapy
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment
Procedure: stress management therapy

SUMMARY:
RATIONALE: Mindful movement is a self-directed activity of mindfulness (intention, attention, and attitude) and physical movement. A mindful movement program may be effective in improving well-being in older women who are breast cancer survivors.

PURPOSE: This randomized clinical trial is studying how well a mindful movement program works in improving quality of life in older female breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the effects of the 12-week Mindful Movement Program on quality of life in older female breast cancer survivors.
* To test the effects of this program on mindfulness outcomes in these participants.
* To compare mindfulness qualities in the experimental group with the control group.
* To determine the qualitative benefits of this program as described by these participants.

OUTLINE: Participants are randomized to 1 of 2 intervention arms.

* Arm I (Mindful Movement Program [MMP]): Participants undergo a 2-hour MMP session once weekly for 12 weeks. Participants are encouraged to practice intentional-mindful movement at home 5 minutes daily during weeks 1-4, 10 minutes daily during weeks 5-8, and 15 minutes daily during weeks 9-12. Mindful movement is a self-directed activity incorporating mindfulness concepts and physical movement. Mindfulness consists of the three core elements: intention (reasons for participating in a mindfulness intervention), attention (observing experiences in the present moment), and attitude (nonjudgmental openness and acceptance of experiences). Each MMP session includes verbal sharing with a partner and the group and movement individually and with a partner, while focusing on the elements of mindfulness. Music is incorporated into some portion of each session.
* Arm II (control): Participants undergo no intervention. All participants complete questionnaires for sociodemographic and individual characteristics, quality of life (including psychological, social, spiritual, and physical well-being, anxiety and depression, fear of recurrence, body image, and upper body symptoms), movement, and mindfulness (including attention, self-compassion, and intention) at baseline and weeks 12 and 18.

PROJECTED ACCRUAL: A total of 75 participants (45 in the experimental group and 30 in the control group) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Breast cancer survivor

  * At least 12 months since completion of treatment (chemotherapy, biotherapy [e.g., trastuzumab], or radiotherapy)
* No evidence of metastatic disease

PATIENT CHARACTERISTICS:

* English speaking
* Not under acute psychological distress
* Not using an assistive device (cane, walker, or wheelchair)
* Able to participate in the Mindful Movement Program by a medical release from the patient's physician
* Pregnancy allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent selective estrogen-receptor modulator permitted
* No other concurrent treatment

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Effects of the Mindful Movement Program on psychological well-being, distress, fear of recurrence, physical well-being, upper-body symptom bother, social well-being, body image, and spiritual well-being at baseline and weeks 12 and 18 | 6 months after study entry
Effects of this program on attention and attitude | 6 months after study entry
Differences of attention and attitude between the experimental group and the control group | 6 months after study entry
Perceptions of the program as described by the experimental group | 6 months after entry

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Crane-Okada, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States